CLINICAL TRIAL: NCT03233308
Title: A Double-Masked, Randomized, Placebo-Controlled Study of Trabecular Outflow Facility Following Treatment With Netarsudil Ophthalmic Solution 0.02% (AR-13324) in Subjects With Elevated Intraocular Pressure
Brief Title: Study of Netarsudil Ophthalmic Solution in Subjects With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-13324-CS206
Record Dates: First submitted 2017-07-12; First posted 2017-07-28 (Actual); Results first posted 2019-06-11 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Primary Open Angle Glaucoma or Ocular Hypertension
Keywords: Aqueous Humor Dynamics; Trabecular Outflow; Netarsudil
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Paired comparison study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Netarsudil Ophthalmic Solution 0.02% (Experimental): Netarsudil Ophthalmic Solution 0.02% was administered in one eye and Placebo comparator in contralateral eye
  Interventions: Drug: Netarsudil Ophthalmic Solution 0.02%; Other: Placebo Comparator
- Placebo Comparator (Placebo Comparator): Placebo comparator administered in one eye and Netarsudil Ophthalmic Solution 0.02% in contralateral eye
  Interventions: Drug: Netarsudil Ophthalmic Solution 0.02%; Other: Placebo Comparator

INTERVENTIONS:
Drug: Netarsudil Ophthalmic Solution 0.02% — 1 drop daily (QD), in the morning (AM) Netarsudil Ophthalmic Solution 0.02% administered to one eye and Placebo comparator to the contralateral eye
Other: Placebo Comparator — 1 drop daily (QD), in the morning (AM) of Placebo comparator administered to one eye and Netarsudil Ophthalmic Solution 0.02% to the contralateral eye

SUMMARY:
To evaluate the effect on trabecular outflow facility of Netarsudil ophthalmic solution 0.02% compared to placebo

DETAILED DESCRIPTION:
Trabecular outflow facility is a measure of aqueous humor dynamics; effect of netarsudil on this parameter as well as on intraocular pressure and episcleral venous pressure was evaluated in this study. Netarsudil treatment was given in one eye and placebo given in contralateral eye for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older
2. Diagnosis of open primary angle glaucoma(POAG) or ocular hypertension (OHT) in both eyes
3. Unmedicated intraocular pressure (IOP) >20 mmHg and < 30 mmHg in both eyes at first qualification visit
4. Best corrected visual acuity (BCVA) equivalent to 20/200 Snellen or better
5. Able to give informed consent and follow study instructions

Exclusion Criteria:

Ophthalmic:

1. Clinically significant ocular disease
2. Pseudoexfoliation or pigment dispersion component glaucoma, history of angle closure glaucoma, or narrow angles
3. Intraocular pressure ≥30 mmHg in either eye
4. A difference in IOP between eyes >4mmHg at qualification visit
5. Use of more than two ocular hypotensive medications within 30 days of screening
6. Known hypersensitivity to any component of the formulation
7. Previous glaucoma surgery or refractive surgery
8. Keratorefractive surgery in either eye
9. Report of ocular injury in either eye within the six months prior to screening or ocular or non-refractive surgery within 3 months prior to screening
10. Recent or current ocular infection or inflammation in either eye
11. Use of ocular medication in either eye of any kind within 30 days of screening
12. Mean central corneal thickness greater than 620 μm in either eye
13. Any abnormality preventing reliable applanation tonometry of either eye
14. Lack of suitable episcleral vein prior to performing Episcleral Venus Pressure (EVP) measurement (applicable to 1 site only)

    Systemic:
15. Clinically significant abnormalities within 6 weeks prior to screening
16. Clinically significant systemic disease
17. Participation in any investigational study within 60 days prior to screening
18. Use of systemic medication that could have an effect on intraocular pressure within 30 days prior to screening
19. Women of childbearing potential who were pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ramirez-Davis, Study Director — Aerie Pharmaceuticals
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Duke Eye Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Randomized Patients: 1 drop daily (QD), in the morning (AM) Netarsudil Ophthalmic Solution 0.02% administered to one eye and Placebo comparator to the contralateral eye
Period: Overall Study
Arm/Group | All Randomized Patients
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population
Arm/Group | All Randomized Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Mean Diurnal Trabecular Outflow Facility
Description: Mean diurnal change from baseline in trabecular (tonographic) outflow facility.
Time Frame: Study treatment was administered for 7 days, and outcome measures collected on Day 8
Population: Modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: mcl/min/mmHg
Groups:
- Netarsudil Ophthalmic Solution 0.02%: Netarsudil Ophthalmic Solution 0.02% was administered in one eye
- Placebo Comparator: Placebo Comparator administered in contralateral eye
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Placebo Comparator
Number analyzed (Participants) | 18 | 18
mcl/min/mmHg | 0.039 (0.0401) | 0.007 (0.0275)
Statistical Analysis 1: Comparison: Netarsudil Ophthalmic Solution 0.02%; Mean Change from Baseline; Test type: Other; p = 0.0010, t-test, 1 sided

2. Primary Outcome: Mean Percent Change From Baseline in the Mean Diurnal Trabecular Outflow Facility.
Description: Mean diurnal change from baseline in trabecular (tonographic) outflow facility.
Time Frame: Study treatment was administered for 7 days, and outcome measures collected on Day 8
Population: Modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Placebo Comparator
Number analyzed (Participants) | 18 | 18
percentage change | 34.589 (34.5935) | 9.597 (25.6334)
Statistical Analysis 1: Comparison: Netarsudil Ophthalmic Solution 0.02%; Mean change from baseline (percent difference from baseline); Test type: Other; p = 0.0003, t-test, 1 sided

3. Secondary Outcome: Mean Change From Baseline in Episcleral Venous Pressure (EVP) and in Intraocular Pressure (IOP)
Description: Mean diurnal change from baseline in mean diurnal IOP measured using a Pneumatonometer and mean diurnal EVP using a custom-modified slit-lamp mounted venomanometer. (EVP conducted at a single site in only 9 participants)
Time Frame: Study treatment was administered for 7 days, and outcome measures collected on Day 8
Population: Modified intent-to-treat (mITT) population, EVP analyzed in 9 participants
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Netarsudil Ophthalmic Solution 0.02%: Netarsudil Ophthalmic Solution 0.02% administered to one eye and placebo to the contralateral eye
- Placebo Comparator: Placebo Comparator administered to one eye and Netarsudil Ophthalmic Solution 0.02% to the contralateral eye
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Placebo Comparator
Number analyzed (Participants) | 18 | 18
mmHg
  Diurnal EVP (delta vs.baseline): number analyzed (Participants) | 9 | 9
  Diurnal EVP (delta vs.baseline) | -0.787 (0.8372) | 0.103 (0.7094)
  Diurnal IOP (delta vs.baseline) | -4.521 (1.5842) | -0.979 (1.6009)
Statistical Analysis 1: Comparison: Netarsudil Ophthalmic Solution 0.02%; Mean change from baseline -EVP; Test type: Other; p = 0.0687, t-test, 1 sided
Statistical Analysis 2: Comparison: Netarsudil Ophthalmic Solution 0.02%; Mean change from baseline -IOP; Test type: Other; p < 0.0001, t-test, 1 sided

4. Secondary Outcome: Mean Percent Change From Baseline in Episcleral Venous Pressure (EVP) and in Intraocular Pressure (IOP)
Description: as for outcome 3
Time Frame: Study treatment was administered for 7 days, and outcome measures collected on Day 8
Population: Modified intent-to-treat (mITT) population, EVP analyzed in 9 participants
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Netarsudil Ophthalmic Solution 0.02%: Netarsudil Ophthalmic Solution 0.02% administered to one eye and Placebo comparator to the contralateral eye
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Placebo Comparator
Number analyzed (Participants) | 18 | 18
percentage change
  Percent change from baseline (EVP): number analyzed (Participants) | 9 | 9
  Percent change from baseline (EVP) | -9.465 (9.5044) | 3.103 (7.7322)
  Percent change from baseline (IOP) | -19.568 (6.0713) | -4.227 (6.9699)
Statistical Analysis 1: Comparison: Netarsudil Ophthalmic Solution 0.02%; Mean change from baseline (percent difference from baseline) -EVP; Test type: Other; p = 0.0087, t-test, 1 sided
Statistical Analysis 2: Comparison: Netarsudil Ophthalmic Solution 0.02%; Mean change from baseline (percent difference from baseline)- IOP; Test type: Other; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 7 Days
Groups:
- Placebo Comparator: Placebo comparator was administered in one eye and Netarsudil Ophthalmic Solution 0.02% in contralateral eye
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 13/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil Ophthalmic Solution 0.02% (N=20) | Placebo Comparator (N=20)
Conjunctival Hyperaemia (Eye disorders) | 13 (13) | 0 (0)
Eye Irritation (Eye disorders) | 3 (3) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 0 (0)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT03233308/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03233308/SAP_001.pdf